CLINICAL TRIAL: NCT04389073
Title: Safety and Efficacy of Metronomic Vinorelbine in Combination With Toripalimab for Patients With HER2- Metastatic Breast Cancer
Brief Title: Safety and Efficacy of Toripalimab in HER2- Metastatic Breast Cancer Patients Treated With Metronomic Vinorelbine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Huanxing Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2167
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; toripalimab; Bevacizumab; Cyclophosphamide; Capecitabine; Tablets; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1 (PD-1+NVB) (Experimental): The treatments received are:
  * Vinorelbine (40 mg/day, tiw, per os)
  * Toripalimab (240 mg every 3 weeks, intravenously [IV]).
  Interventions: Drug: Vinorelbine 40mg; Biological: Toripalimab 240mg
- Arm 2 (PD-1+NVB+Bev) (Experimental): The treatments received are:
  * Vinorelbine (40 mg/day, tiw, per os)
  * Toripalimab (240 mg every 3 weeks, intravenously [IV])
  * Bevacizumab (5 mg/kg every 3 weeks, intravenously [IV]).
  Interventions: Drug: Vinorelbine 40mg; Biological: Toripalimab 240mg; Biological: Bevacizumab 5 mg/kg
- Arm 3 (PD-1+NVB+DDP) (Experimental): * Vinorelbine (40 mg/day, tiw, per os)
  * Toripalimab (240 mg every 3 weeks, intravenously [IV])
  * Cisplatin (50mg/m2 every 3 weeks, intravenously [IV]).
  Interventions: Drug: Vinorelbine 40mg; Biological: Toripalimab 240mg; Drug: Cisplatin
- Arm 4 (PD-1+VEX) (Experimental): * Vinorelbine (40 mg/day, tiw, per os)
  * Toripalimab (240 mg every 3 weeks, intravenously [IV])
  * Cyclophosphamide (50 mg/day, qd, per os)
  * Capecitabine (500 mg, tid, per os)
  Interventions: Drug: Vinorelbine 40mg; Biological: Toripalimab 240mg; Drug: Cyclophosphamide 50 mg; Drug: Capecitabine 500Mg Oral Tablet
- Arm 5 (NVB) (Active Comparator): • Vinorelbine (40 mg/day, tiw, per os)
  Interventions: Drug: Vinorelbine 40mg

INTERVENTIONS:
Drug: Vinorelbine 40mg — Two tablets per day, three times a week. Vinorelbine will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
Biological: Toripalimab 240mg — Toripalimab 240 MG IV infusion every 3 weeks. Toripalimab will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Other Names: JS001
  Arms: Arm 1 (PD-1+NVB); Arm 2 (PD-1+NVB+Bev); Arm 3 (PD-1+NVB+DDP); Arm 4 (PD-1+VEX)
Biological: Bevacizumab 5 mg/kg — Bevacizumab 5 mg/kg IV infusion every 3 weeks. Bevacizumab will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Arms: Arm 2 (PD-1+NVB+Bev)
Drug: Cyclophosphamide 50 mg — 50 mg per day. Cyclophosphamide will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Arms: Arm 4 (PD-1+VEX)
Drug: Capecitabine 500Mg Oral Tablet — 500mg three times a day. Capecitabine will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Arms: Arm 4 (PD-1+VEX)
Drug: Cisplatin — Cisplatin 50mg/m2 IV infusion every 3 weeks. Cisplatin will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Arms: Arm 3 (PD-1+NVB+DDP)

SUMMARY:
The investigators hypothesize that the administration of Toripalimab (anti-PD-1 antibody, JS001) combined to metronomic Vinorelbine may be an interesting therapeutic option for female patients with HER2- metastatic breast cancer. The approach suggested here is to deplete and active the immune response of these patients. The combination of Toripalimab and Vinorelbine would provide a higher gain in anti-tumor response in these patients than in those with chemotherapy alone.

The investigators proposal is to conduct a multicentric, single arm, Phase II trial in HER2- patients with metastatic breast cancer, aiming to evaluate the clinical activity of the combination therapy Toripalimab + metronomic Vinorelbine. Patients will receive Vinorelbine (40 mg/day, tiw, per os) and Toripalimab (240 mg every 3 weeks, intravenously [IV]). The adverse events of the two drugs are well known.

DETAILED DESCRIPTION:
Both study drugs will continue to be administered as long as patient experience clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with life expectancy ≥ 3 months, age ≥ 18 years at the time
* informed consent is signed.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 as assessed within 21 days prior to first dosage.
* Subjects with HER2 negative metastasis breast cancer, source documented, defined as per American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) guidelines.
* Subjects previously treated with no more than one prior line of standard chemotherapy
* Subjects with measurable metastatic disease defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) guidelines.
* Subjects may previously exposed to anthracyclines (e.g. doxorubicin, epirubicin) and/or taxanes (e.g., paclitaxel, docetaxel) including:

  * has been pretreated in the adjuvant or neoadjuvant setting with anthracyclines and/or taxanes before breast cancer relapsing;
  * has experienced treatment failure while receiving or after completing anthracycline- and/or taxane- based chemotherapy;
  * not suitable for the choice of anthracycline- and/or taxane- based chemotherapy as first-line treatment in the judgment of investigator.
* Prior radiotherapy must have completed before randomization, with full recovery from acute radiation side effects. An interval of less than 4 weeks after radiotherapy was not allowed.Concurrent limited field radiation therapy (RT) is allowed. At least one measurable lesion must be completely outside the radiation portal in accordance with RECIST 1.1 guidelines;
* At least 30 days from major surgery before randomization, with full recovery;
* Adequate bone marrow function as evidenced by the following:

  * Absolute Neutrophil Count (ANC) ≥ 1500/mm2;
  * Platelets ≥ 100,000/mm2;
  * Hemoglobin (Hb) ≥ 10 g/dL.
* Adequate liver function as evidenced by the following:

  * Total serum bilirubin ≤ 1.5 times upper limit of normal range (ULN);
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 times ULN (if hepatic metastases present ≤ 5.0 times ULN);
  * Alkaline phosphatase < 5 x ULN.
* Adequate renal function as evidenced by the following:

  * Creatinine clearance > 40 mL/min (by Cockcroft-Gault).
* Women of child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of randomization and agree to take an adequate contraceptive measure.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* History of, or current active cancer other than breast cancer, with the exception of curatively resected non-melanomatous skin cancer, curatively treated cervical carcinoma in situ, or other primary solid tumors curatively treated with no known active disease present and no curative treatment administered for the last 3 years.
* Patients with medical conditions that the only manifestation is hydrothorax, ascites, bone lesions or other un-measurable diseases.
* Subjects with visceral crisis in the judgment of investigator. Visceral crisis is defined as severe organ dysfunction as assessed by signs and symptoms, laboratory studies, and rapid progression of disease. Visceral crisis is not the mere presence of disease of visceral metastases, but implies important visceral compromise leading to a clinical indication for a more rapidly efficacious therapy, particularly since chemotherapy option at progression will probably not be possible.
* Malabsorption syndrome or disease significantly affecting gastro-intestinal function or major resection of the stomach or proximal small bowel that could affect absorption of Oral NVB.
* Subjects with dysphagia, or inability to swallow the tablets.
* Subjects with symptoms suggesting central nervous system (CNS) involvement or leptomeningeal metastases, any suspicious sins or symptoms of CNS involvement or leptomeningeal metastases should be excluded by CT or MRI scans.
* Other serious illness or medical conditions by the investigator during screening:

  * Clinically significant cardiac disease;
  * Unstable diabetes;
  * Uncontrolled hypercalcemia;
  * Clinically significant active infections (current or in the last two weeks).
* Previous organ allograft.
* Current peripheral neuropathy ≥grade 2 according to NCI version 4.0 criteria.
* Concomitant hormonal therapy for MBC.
* Ongoing anti-coagulation therapy.
* Subjects of reproductive potential who are pregnant, breast feeding or not willing to use effective contraceptive precautions during the study and for at least one month after the last dose of investigational product in the judgment of the investigator.
* Patients with psychiatric disorder or other disease leading to incompliance to the therapy.
* An interval of less than 3 weeks between the last dose of previous chemotherapy and randomization.
* Previous treated by oral NVB.
* Treatment with any investigational drug within 30 days before the beginning of treatment with study drug. Less than 30 days since receipt of any other investigational product or device.
* Known hypersensitivity to any ingredient of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 6 weeks of treatment
  CBR, defined as the percentage of Complete Response (CR), (Partial Response) PR or Stable Disease (SD) . Response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) V1.1.

SECONDARY OUTCOMES:
Overall response Rate (ORR) | 6 weeks of treatment
  The objective response rate (ORR) will be defined as the proportion of patients (described on the efficacy-evaluable population) who achieve complete response (CR) or partial response (PR) as best overall response at 6 weeks of treatment. ORR is based on tumor assessments.
Progression-Free Survival (PFS) | 15 months
  Measured from the date of study drugs start to the date of the first objective disease progression or death.
Overall Survival (OS) | 15 months
  Defined as the duration of time from start of treatment to time of death.
Adverse events reporting | 15 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Huanxing Cancer Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Mo H, Yu Y, Sun X, Ge H, Yu L, Guan X, Zhai J, Zhu A, Wei Y, Wang J, Yan X, Qian H, Xu B, Ma F. Metronomic chemotherapy plus anti-PD-1 in metastatic breast cancer: a Bayesian adaptive randomized phase 2 trial. Nat Med. 2024 Sep;30(9):2528-2539. doi: 10.1038/s41591-024-03088-2. Epub 2024 Jul 5. PMID 38969879